CLINICAL TRIAL: NCT03192995
Title: Treatment With Lorcaserin for Cocaine Use: The TLC Study
Acronym: TLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA alert regarding study drug safety
Sponsor: Glenn-Milo Santos (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Glenn-Milo Santos, Senior Research Scientist, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-21502; 1R34DA042161 (NIH)
Record Dates: First submitted 2017-06-12; First posted 2017-06-20 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cocaine Use Disorder
Keywords: HIV; sexual behavior
MeSH Terms: conditions — Sexual Behavior | interventions — lorcaserin; Ecological Momentary Assessment

STUDY DESIGN:
Intervention Model Description: 12-week parallel group pilot study with 2:1 random assignment to 20 mg of extended-release oral lorcaserin versus placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): lorcaserin, extended release, Substance use counseling, ACASI behavioral questionnaire, BART, and ecological momentary assessment
  Interventions: Drug: lorcaserin; Behavioral: Substance use counseling; Behavioral: ACASI; Diagnostic Test: Cocaine metabolites; Behavioral: Ecological Momentary Assessment (EMA); Behavioral: Balloon Analogue Risk Task (BART); Behavioral: Qualitative Exit Interview
- Control (Placebo Comparator): Placebo, Substance use counseling, ACASI behavioral questionnaire, BART, and ecological momentary assessment
  Interventions: Drug: Placebo Oral Tablet; Behavioral: Substance use counseling; Behavioral: ACASI; Diagnostic Test: Cocaine metabolites; Behavioral: Ecological Momentary Assessment (EMA); Behavioral: Balloon Analogue Risk Task (BART); Behavioral: Qualitative Exit Interview

INTERVENTIONS:
Drug: lorcaserin — lorcaserin 20 mg tablet
  Other Names: BELVIQ
  Arms: Experimental
Drug: Placebo Oral Tablet — placebo 20 mg. tablet
  Other Names: Placebo
  Arms: Control
Behavioral: Substance use counseling — Manual-driven psychosocial substance use counseling program using cognitive behavioral therapy and motivational interviewing techniques and incorporating the Stages of Change Model.
Behavioral: ACASI — Audio-computer assisted self-interviews (ACASI) is a self-administered standardized questionnaire on substance and alcohol use, substance use treatment, sexual risk behavior, partnership sexual risk, and
Diagnostic Test: Cocaine metabolites — Rapid qualitative urine test Medtox Verdict II (Medtox Diagnostics, Burlington, NC) and tamper-evident sweat patches (PharmChek®, PharmChem, Inc., Fort Worth, Tx)
Behavioral: Ecological Momentary Assessment (EMA) — EMA are questions sent to the participant 4-5 times a day to determine real-time behavior and participant experiences.
  Other Names: EMA
Behavioral: Balloon Analogue Risk Task (BART) — BART is a computerized measure of risk taking behavior. The BART models real-world risk behavior through the conceptual frame of balancing the potential for reward versus loss. This is a test for impulsivity.
  Other Names: BART
Behavioral: Qualitative Exit Interview — The qualitative exit interview assessed acceptability measures and included questions on attitudes about trial participation, level of satisfaction with trial procedures, and trial medication.

SUMMARY:
This project is a placebo-controlled, double-blind randomized trial evaluating the feasibility, tolerability, acceptability and adherence for lorcaserin among actively using, men who have sex with men (MSM) with cocaine use disorders.The study will enroll 45 individuals who will randomly be assigned to either the treatment (lorcaserin) arm or the placebo arm, to be taken twice a day for 12 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 12-week parallel group pilot study with 2:1 random assignment to 20 mg of extended-release oral lorcaserin versus placebo. Participants are recruited via street outreach, recruitment flyers, sexually transmitted diseases (STD) and HIV clinics, needle exchanges, community organizations, MSM bars, online Web sites, and social media. Potential participants complete a brief telephone screen to assess initial eligibility and, if eligible, are scheduled for an in-person screening visit. All participants give informed consent using University of California at San Francisco (UCSF) Institutional Review Board (IRB)-approved consent forms. A 10-item true/false questionnaire is used to verify participants' understanding of the trial. The target sample size for the study was 45 participants (The Food and Drug Administration (FDA) closed down the study early due to a long-term safety study showing that long term use of lorcaserin could be hazardous to your health). Only 22 of the 45 participants were randomized to the study.

With the proposed sample size, we estimate that proportions for our feasibility and acceptability outcomes would be estimated within margins of sampling error (Mean squared error (MSEs); i.e., half widths of 95% confidence intervals) of ≤14.4 percentage points, and means with MSEs of 0.30 standard deviations, both typical for a small pilot study.

Participants are screened for eligibility based on inclusion criteria. At Enrollment, participants are instructed to take one pill each day of extended-release lorcaserin 20mg or placebo. Medications are dispensed in bottles with Medication Events Monitoring (MEMS) caps, which are wireless medication monitoring devices that record each opening as a real-time medication event. All participants are asked about potential adverse events at each follow-up visit; symptom-driven physical exams and safety laboratory monitoring are done at weeks 4, 8, and 12. Adverse events are classified using the Division of AIDS (DAIDS) Table for Grading Severity of Adult Adverse Experiences for HIV Prevention Trials Network. Participants are seen every week for substance use counseling and urine tests for cocaine metabolites. Trained staff, supervised by a clinical psychologist, administered brief (20-30 minutes) substance use counseling at follow-up visits. Audio-computer assisted self-interviews (ACASI) are used to standardize data collection and minimize reporting bias. Standardized measures are used to assess drug and alcohol use using timeline followback, substance use treatment, craving and severity of cocaine dependence, and sexual risk behavior. Acceptability measures include questions on attitudes about trial participation, level of satisfaction with trial procedures, and trial medication.

ELIGIBILITY:
Inclusion Criteria:

* Male gender assigned at birth and transgender men;
* self-reported anal intercourse with men in the prior six months while under the influence of cocaine;
* cocaine use disorder by (Diagnostic and Statistical Manual of Mental Health Disorders (DSM-V) and Structured clinical interviews (SCID) criteria;
* current cocaine use confirmed by urinalysis and cocaine use at least 15 days in the past 30 days;
* HIV-negative by rapid test or HIV-positive with a medical record of HIV infection;
* no current acute illnesses requiring prolonged medical care;
* no chronic illnesses that are likely to progress clinically during trial;
* able and willing to provide informed consent and adhere to visit schedule;
* age 18-65 years;
* baseline complete blood count (CBC), total protein, albumin, glucose, alkaline phosphatase, creatinine, Blood Urea Nitrogen (BUN), and electrolytes without clinically significant abnormalities as determined by study clinician in conjunction with symptoms, physical exam, and medical history

Exclusion Criteria:

* Any psychiatric condition (e.g., depression with suicidal ideation, schizophrenia) or medical condition that would preclude safe study participation;
* HIV-positive test result at screening visit but previously unaware of HIV infection (i.e., newly diagnosed with HIV infection at screening; those with a medical record of HIV infection are eligible);
* any moderate to severe alcohol or substance use disorders (other than cocaine use disorders), according to DSM-V criteria;
* known allergy or previous adverse reaction to lorcaserin;
* current T-cell count (CD4) count < 200 cells/mm3 ;
* moderate/sever liver disease (Aspartate Transferase (AST), Alanine Transaminase (ALT) > 3 times upper limit or normal);
* severely impaired renal function (creatinine clearance £ 30 ml/min);
* use of medications that affect the serotonergic neurotransmitter system (e.g., selective serotonin reuptake inhibitors (SSRIs), selective serotonin-norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, monoamine oxidase inhibitors (MAOIs));
* predisposition to priapism;
* currently participating in another longitudinal intervention research study;
* body mass index (BMI) < 15; or ≥ 30 with desire to use weight management medication, or BMI > 35;
* anticipated use of agents that are associated with valvulopathy and/or pulmonary hypertension
* Are currently treated with an opiate-substitute (buprenorphine or methadone) maintenance treatment or received therapy with any opiate-substitute within 30 days preceding screening
* Currently in court-mandated cocaine use treatment;
* Had previous history of suicidal behavior in the last 12 months ("yes" answer to the suicidal behavior question 6 of the Columbia-Suicide Severity Rating Scale (C-SSRS)); or currently have suicidal ideation as determined by 'yes' answers to questions 4 or 5 on the C-SSRS administered by a study clinician;
* Any physical condition affecting drug absorption (e.g., gastrectomy);
* 12-lead Electrocardiogram (ECG) demonstrating Corrected QT interval (QTc) > 450 or a Q wave, R wave and S wave (QRS) interval > 120 msec at screening. If Fridericia (QTcF) exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility.

(Note: Participants newly diagnosed with HIV at screening who consent to be contacted for re-screening will be called in the subsequent month, or later, depending on participant preference).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn-Milo Santos, PhD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Department of Public Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riezzo I, Fiore C, De Carlo D, Pascale N, Neri M, Turillazzi E, Fineschi V. Side effects of cocaine abuse: multiorgan toxicity and pathological consequences. Curr Med Chem. 2012;19(33):5624-46. doi: 10.2174/092986712803988893. PMID 22934772
- [Background] Karila L, Petit A, Lowenstein W, Reynaud M. Diagnosis and consequences of cocaine addiction. Curr Med Chem. 2012;19(33):5612-8. doi: 10.2174/092986712803988839. PMID 22856661
- [Background] Crane EH. Highlights of the 2011 Drug Abuse Warning Network (DAWN) Findings on Drug-Related Emergency Department Visits. 2013 Feb 22. In: The CBHSQ Report. Rockville (MD): Substance Abuse and Mental Health Services Administration (US); 2013-. Available from http://www.ncbi.nlm.nih.gov/books/NBK384680/ PMID 27631059
- [Background] Degenhardt L, Baxter AJ, Lee YY, Hall W, Sara GE, Johns N, Flaxman A, Whiteford HA, Vos T. The global epidemiology and burden of psychostimulant dependence: findings from the Global Burden of Disease Study 2010. Drug Alcohol Depend. 2014 Apr 1;137:36-47. doi: 10.1016/j.drugalcdep.2013.12.025. Epub 2014 Jan 27. PMID 24559607
- [Background] Vandhuick O, Pistorius MA, Jousse S, Ferreira-Maldent N, Guilmot JL, Guias B, Bressollette L. [Drug addiction and cardiovascular pathologies]. J Mal Vasc. 2004 Dec;29(5):243-8. doi: 10.1016/s0398-0499(04)96768-6. French. PMID 15738835
- [Background] Kloner RA, Hale S, Alker K, Rezkalla S. The effects of acute and chronic cocaine use on the heart. Circulation. 1992 Feb;85(2):407-19. doi: 10.1161/01.cir.85.2.407. PMID 1346509
- [Background] McCord J, Jneid H, Hollander JE, de Lemos JA, Cercek B, Hsue P, Gibler WB, Ohman EM, Drew B, Philippides G, Newby LK; American Heart Association Acute Cardiac Care Committee of the Council on Clinical Cardiology. Management of cocaine-associated chest pain and myocardial infarction: a scientific statement from the American Heart Association Acute Cardiac Care Committee of the Council on Clinical Cardiology. Circulation. 2008 Apr 8;117(14):1897-907. doi: 10.1161/CIRCULATIONAHA.107.188950. Epub 2008 Mar 17. No abstract available. PMID 18347214
- [Background] Phillips K, Luk A, Soor GS, Abraham JR, Leong S, Butany J. Cocaine cardiotoxicity: a review of the pathophysiology, pathology, and treatment options. Am J Cardiovasc Drugs. 2009;9(3):177-96. doi: 10.2165/00129784-200909030-00005. PMID 19463023
- [Background] Steinhauer JR, Caulfield JB. Spontaneous coronary artery dissection associated with cocaine use: a case report and brief review. Cardiovasc Pathol. 2001 May-Jun;10(3):141-5. doi: 10.1016/s1054-8807(01)00074-6. PMID 11485859
- [Background] Sanchez T, Finlayson T, Drake A, Behel S, Cribbin M, Dinenno E, Hall T, Kramer S, Lansky A; Centers for Disease Control and Prevention (CDC). Human immunodeficiency virus (HIV) risk, prevention, and testing behaviors--United States, National HIV Behavioral Surveillance System: men who have sex with men, November 2003-April 2005. MMWR Surveill Summ. 2006 Jul 7;55(6):1-16. PMID 16826162
- [Background] Raymond HF, Chen YH, Ick T, Scheer S, Bernstein K, Liska S, Louie B, Pandori M, McFarland W. A new trend in the HIV epidemic among men who have sex with men, San Francisco, 2004-2011. J Acquir Immune Defic Syndr. 2013 Apr 15;62(5):584-9. doi: 10.1097/QAI.0b013e318285febf. PMID 23334505
- [Background] Mimiaga MJ, Reisner SL, Fontaine YM, Bland SE, Driscoll MA, Isenberg D, Cranston K, Skeer MR, Mayer KH. Walking the line: stimulant use during sex and HIV risk behavior among Black urban MSM. Drug Alcohol Depend. 2010 Jul 1;110(1-2):30-7. doi: 10.1016/j.drugalcdep.2010.01.017. Epub 2010 Mar 23. PMID 20334986
- [Background] Colfax G, Vittinghoff E, Husnik MJ, McKirnan D, Buchbinder S, Koblin B, Celum C, Chesney M, Huang Y, Mayer K, Bozeman S, Judson FN, Bryant KJ, Coates TJ; EXPLORE Study Team. Substance use and sexual risk: a participant- and episode-level analysis among a cohort of men who have sex with men. Am J Epidemiol. 2004 May 15;159(10):1002-12. doi: 10.1093/aje/kwh135. PMID 15128613
- [Background] Ober A, Shoptaw S, Wang PC, Gorbach P, Weiss RE. Factors associated with event-level stimulant use during sex in a sample of older, low-income men who have sex with men in Los Angeles. Drug Alcohol Depend. 2009 Jun 1;102(1-3):123-9. doi: 10.1016/j.drugalcdep.2009.02.002. Epub 2009 Mar 26. PMID 19327917
- [Background] Mackesy-Amiti ME, Fendrich M, Johnson TP. Symptoms of substance dependence and risky sexual behavior in a probability sample of HIV-negative men who have sex with men in Chicago. Drug Alcohol Depend. 2010 Jul 1;110(1-2):38-43. doi: 10.1016/j.drugalcdep.2010.01.016. Epub 2010 Mar 9. PMID 20219291
- [Background] Lambert G, Cox J, Hottes TS, Tremblay C, Frigault LR, Alary M, Otis J, Remis RS; M-Track Study Group. Correlates of unprotected anal sex at last sexual episode: analysis from a surveillance study of men who have sex with men in Montreal. AIDS Behav. 2011 Apr;15(3):584-95. doi: 10.1007/s10461-009-9605-3. PMID 20033763
- [Background] Bowers JR, Branson CM, Fletcher JB, Reback CJ. Predictors of HIV Sexual Risk Behavior among Men Who Have Sex with Men, Men Who Have Sex with Men and Women, and Transgender Women. Int J Sex Health. 2012;24(4):290-302. doi: 10.1080/19317611.2012.715120. PMID 24660042
- [Background] Santos GM, Coffin PO, Das M, Matheson T, DeMicco E, Raiford JL, Vittinghoff E, Dilley JW, Colfax G, Herbst JH. Dose-response associations between number and frequency of substance use and high-risk sexual behaviors among HIV-negative substance-using men who have sex with men (SUMSM) in San Francisco. J Acquir Immune Defic Syndr. 2013 Aug 1;63(4):540-4. doi: 10.1097/QAI.0b013e318293f10b. PMID 23572012
- [Background] Tyndall MW, Currie S, Spittal P, Li K, Wood E, O'Shaughnessy MV, Schechter MT. Intensive injection cocaine use as the primary risk factor in the Vancouver HIV-1 epidemic. AIDS. 2003 Apr 11;17(6):887-93. doi: 10.1097/00002030-200304110-00014. PMID 12660536
- [Background] Cepeda JA, Vickerman P, Bruneau J, Zang G, Borquez A, Farrell M, Degenhardt L, Martin NK. Estimating the contribution of stimulant injection to HIV and HCV epidemics among people who inject drugs and implications for harm reduction: A modeling analysis. Drug Alcohol Depend. 2020 Aug 1;213:108135. doi: 10.1016/j.drugalcdep.2020.108135. Epub 2020 Jun 24. PMID 32603976
- [Background] Ostrow DG, Plankey MW, Cox C, Li X, Shoptaw S, Jacobson LP, Stall RC. Specific sex drug combinations contribute to the majority of recent HIV seroconversions among MSM in the MACS. J Acquir Immune Defic Syndr. 2009 Jul 1;51(3):349-55. doi: 10.1097/QAI.0b013e3181a24b20. PMID 19387357
- [Background] Koblin BA, Husnik MJ, Colfax G, Huang Y, Madison M, Mayer K, Barresi PJ, Coates TJ, Chesney MA, Buchbinder S. Risk factors for HIV infection among men who have sex with men. AIDS. 2006 Mar 21;20(5):731-9. doi: 10.1097/01.aids.0000216374.61442.55. PMID 16514304
- [Background] Ostrow DG, DiFranceisco WJ, Chmiel JS, Wagstaff DA, Wesch J. A case-control study of human immunodeficiency virus type 1 seroconversion and risk-related behaviors in the Chicago MACS/CCS Cohort, 1984-1992. Multicenter AIDS Cohort Study. Coping and Change Study. Am J Epidemiol. 1995 Oct 15;142(8):875-83. doi: 10.1093/oxfordjournals.aje.a117727. PMID 7572964
- [Background] Hinkin CH, Barclay TR, Castellon SA, Levine AJ, Durvasula RS, Marion SD, Myers HF, Longshore D. Drug use and medication adherence among HIV-1 infected individuals. AIDS Behav. 2007 Mar;11(2):185-94. doi: 10.1007/s10461-006-9152-0. PMID 16897351
- [Background] Carrico AW. Substance use and HIV disease progression in the HAART era: implications for the primary prevention of HIV. Life Sci. 2011 May 23;88(21-22):940-7. doi: 10.1016/j.lfs.2010.10.002. Epub 2010 Oct 8. PMID 20934437
- [Background] Shoptaw S, Stall R, Bordon J, Kao U, Cox C, Li X, Ostrow DG, Plankey MW. Cumulative exposure to stimulants and immune function outcomes among HIV-positive and HIV-negative men in the Multicenter AIDS Cohort Study. Int J STD AIDS. 2012 Aug;23(8):576-80. doi: 10.1258/ijsa.2012.011322. PMID 22930295
- [Background] Cook JA, Burke-Miller JK, Cohen MH, Cook RL, Vlahov D, Wilson TE, Golub ET, Schwartz RM, Howard AA, Ponath C, Plankey MW, Levine AM, Grey DD. Crack cocaine, disease progression, and mortality in a multicenter cohort of HIV-1 positive women. AIDS. 2008 Jul 11;22(11):1355-63. doi: 10.1097/QAD.0b013e32830507f2. PMID 18580615
- [Background] Chan B, Kondo K, Freeman M, Ayers C, Montgomery J, Kansagara D. Pharmacotherapy for Cocaine Use Disorder-a Systematic Review and Meta-analysis. J Gen Intern Med. 2019 Dec;34(12):2858-2873. doi: 10.1007/s11606-019-05074-8. Epub 2019 Jun 10. PMID 31183685
- [Background] Higgins GA, Fletcher PJ, Shanahan WR. Lorcaserin: A review of its preclinical and clinical pharmacology and therapeutic potential. Pharmacol Ther. 2020 Jan;205:107417. doi: 10.1016/j.pharmthera.2019.107417. Epub 2019 Oct 16. PMID 31629010
- [Background] Rothman RB, Blough BE, Baumann MH. Dopamine/serotonin releasers as medications for stimulant addictions. Prog Brain Res. 2008;172:385-406. doi: 10.1016/S0079-6123(08)00919-9. PMID 18772043
- [Background] Higgins GA, Sellers EM, Fletcher PJ. From obesity to substance abuse: therapeutic opportunities for 5-HT2C receptor agonists. Trends Pharmacol Sci. 2013 Oct;34(10):560-70. doi: 10.1016/j.tips.2013.08.001. Epub 2013 Sep 13. PMID 24041919
- [Background] Alex KD, Pehek EA. Pharmacologic mechanisms of serotonergic regulation of dopamine neurotransmission. Pharmacol Ther. 2007 Feb;113(2):296-320. doi: 10.1016/j.pharmthera.2006.08.004. Epub 2006 Oct 17. PMID 17049611
- [Background] Bubar MJ, Cunningham KA. Serotonin 5-HT2A and 5-HT2C receptors as potential targets for modulation of psychostimulant use and dependence. Curr Top Med Chem. 2006;6(18):1971-85. doi: 10.2174/156802606778522131. PMID 17017968
- [Background] Bubar MJ, Cunningham KA. Prospects for serotonin 5-HT2R pharmacotherapy in psychostimulant abuse. Prog Brain Res. 2008;172:319-46. doi: 10.1016/S0079-6123(08)00916-3. PMID 18772040
- [Background] Burton CL, Rizos Z, Diwan M, Nobrega JN, Fletcher PJ. Antagonizing 5-HT(2)A receptors with M100907 and stimulating 5-HT(2)C receptors with Ro60-0175 blocks cocaine-induced locomotion and zif268 mRNA expression in Sprague-Dawley rats. Behav Brain Res. 2013 Mar 1;240:171-81. doi: 10.1016/j.bbr.2012.11.030. Epub 2012 Nov 28. PMID 23201361
- [Background] Craige CP, Unterwald EM. Serotonin (2C) receptor regulation of cocaine-induced conditioned place preference and locomotor sensitization. Behav Brain Res. 2013 Feb 1;238:206-10. doi: 10.1016/j.bbr.2012.10.034. Epub 2012 Oct 26. PMID 23103406
- [Background] Cunningham KA, Fox RG, Anastasio NC, Bubar MJ, Stutz SJ, Moeller FG, Gilbertson SR, Rosenzweig-Lipson S. Selective serotonin 5-HT(2C) receptor activation suppresses the reinforcing efficacy of cocaine and sucrose but differentially affects the incentive-salience value of cocaine- vs. sucrose-associated cues. Neuropharmacology. 2011 Sep;61(3):513-23. doi: 10.1016/j.neuropharm.2011.04.034. Epub 2011 May 11. PMID 21575646
- [Background] Filip M, Alenina N, Bader M, Przegalinski E. Behavioral evidence for the significance of serotoninergic (5-HT) receptors in cocaine addiction. Addict Biol. 2010 Jul;15(3):227-49. doi: 10.1111/j.1369-1600.2010.00214.x. Epub 2010 Apr 29. PMID 20456287
- [Background] Filip M, Spampinato U, McCreary AC, Przegalinski E. Pharmacological and genetic interventions in serotonin (5-HT)(2C) receptors to alter drug abuse and dependence processes. Brain Res. 2012 Oct 2;1476:132-53. doi: 10.1016/j.brainres.2012.03.035. Epub 2012 Mar 23. PMID 22494568
- [Background] Katsidoni V, Apazoglou K, Panagis G. Role of serotonin 5-HT2A and 5-HT2C receptors on brain stimulation reward and the reward-facilitating effect of cocaine. Psychopharmacology (Berl). 2011 Feb;213(2-3):337-54. doi: 10.1007/s00213-010-1887-7. Epub 2010 Jun 25. PMID 20577718
- [Background] Leggio GM, Cathala A, Moison D, Cunningham KA, Piazza PV, Spampinato U. Serotonin2C receptors in the medial prefrontal cortex facilitate cocaine-induced dopamine release in the rat nucleus accumbens. Neuropharmacology. 2009 Feb;56(2):507-13. doi: 10.1016/j.neuropharm.2008.10.005. Epub 2008 Oct 17. PMID 18977370
- [Background] Manvich DF, Kimmel HL, Howell LL. Effects of serotonin 2C receptor agonists on the behavioral and neurochemical effects of cocaine in squirrel monkeys. J Pharmacol Exp Ther. 2012 May;341(2):424-34. doi: 10.1124/jpet.111.186981. Epub 2012 Feb 10. PMID 22328576
- [Background] Pockros LA, Pentkowski NS, Conway SM, Ullman TE, Zwick KR, Neisewander JL. 5-HT(2A) receptor blockade and 5-HT(2C) receptor activation interact to reduce cocaine hyperlocomotion and Fos protein expression in the caudate-putamen. Synapse. 2012 Dec;66(12):989-1001. doi: 10.1002/syn.21592. Epub 2012 Sep 11. PMID 22886755
- [Background] Grottick AJ, Fletcher PJ, Higgins GA. Studies to investigate the role of 5-HT(2C) receptors on cocaine- and food-maintained behavior. J Pharmacol Exp Ther. 2000 Dec;295(3):1183-91. PMID 11082456
- [Background] Pelloux Y, Dilleen R, Economidou D, Theobald D, Everitt BJ. Reduced forebrain serotonin transmission is causally involved in the development of compulsive cocaine seeking in rats. Neuropsychopharmacology. 2012 Oct;37(11):2505-14. doi: 10.1038/npp.2012.111. Epub 2012 Jul 4. PMID 22763621
- [Background] Pirtle JL, Hickman MD, Boinpelly VC, Surineni K, Thakur HK, Grasing KW. The serotonin-2C agonist Lorcaserin delays intravenous choice and modifies the subjective and cardiovascular effects of cocaine: A randomized, controlled human laboratory study. Pharmacol Biochem Behav. 2019 May;180:52-59. doi: 10.1016/j.pbb.2019.02.010. Epub 2019 Feb 24. PMID 30811963
- [Background] Fletcher PJ, Rizos Z, Noble K, Higgins GA. Impulsive action induced by amphetamine, cocaine and MK801 is reduced by 5-HT(2C) receptor stimulation and 5-HT(2A) receptor blockade. Neuropharmacology. 2011 Sep;61(3):468-77. doi: 10.1016/j.neuropharm.2011.02.025. Epub 2011 Mar 21. PMID 21402085
- [Background] Higgins GA, Silenieks LB, Rossmann A, Rizos Z, Noble K, Soko AD, Fletcher PJ. The 5-HT2C receptor agonist lorcaserin reduces nicotine self-administration, discrimination, and reinstatement: relationship to feeding behavior and impulse control. Neuropsychopharmacology. 2012 Apr;37(5):1177-91. doi: 10.1038/npp.2011.303. Epub 2011 Dec 21. PMID 22189292
- [Background] Colfax GN, Santos GM, Das M, Santos DM, Matheson T, Gasper J, Shoptaw S, Vittinghoff E. Mirtazapine to reduce methamphetamine use: a randomized controlled trial. Arch Gen Psychiatry. 2011 Nov;68(11):1168-75. doi: 10.1001/archgenpsychiatry.2011.124. PMID 22065532
- [Background] Bohula EA, Wiviott SD, McGuire DK, Inzucchi SE, Kuder J, Im K, Fanola CL, Qamar A, Brown C, Budaj A, Garcia-Castillo A, Gupta M, Leiter LA, Weissman NJ, White HD, Patel T, Francis B, Miao W, Perdomo C, Dhadda S, Bonaca MP, Ruff CT, Keech AC, Smith SR, Sabatine MS, Scirica BM; CAMELLIA-TIMI 61 Steering Committee and Investigators. Cardiovascular Safety of Lorcaserin in Overweight or Obese Patients. N Engl J Med. 2018 Sep 20;379(12):1107-1117. doi: 10.1056/NEJMoa1808721. Epub 2018 Aug 26. PMID 30145941
- [Background] de Andrade Mesquita L, Fagundes Piccoli G, Richter da Natividade G, Frison Spiazzi B, Colpani V, Gerchman F. Is lorcaserin really associated with increased risk of cancer? A systematic review and meta-analysis. Obes Rev. 2021 Mar;22(3):e13170. doi: 10.1111/obr.13170. Epub 2020 Dec 1. PMID 33258543
- [Background] Centers for Disease Control and Prevention. Revised guidelines for HIV counseling, testing, and referral. MMWR Recomm Rep. 2001 Nov 9;50(RR-19):1-57; quiz CE1-19a1-CE6-19a1. PMID 11718472
- [Background] Haberer JE, Kahane J, Kigozi I, Emenyonu N, Hunt P, Martin J, Bangsberg DR. Real-time adherence monitoring for HIV antiretroviral therapy. AIDS Behav. 2010 Dec;14(6):1340-6. doi: 10.1007/s10461-010-9799-4. PMID 20809380
- [Background] Das M, Santos D, Matheson T, Santos GM, Chu P, Vittinghoff E, Shoptaw S, Colfax GN. Feasibility and acceptability of a phase II randomized pharmacologic intervention for methamphetamine dependence in high-risk men who have sex with men. AIDS. 2010 Apr 24;24(7):991-1000. doi: 10.1097/qad.0b013e328336e98b. PMID 20397286
- [Background] Dunn C, Deroo L, Rivara FP. The use of brief interventions adapted from motivational interviewing across behavioral domains: a systematic review. Addiction. 2001 Dec;96(12):1725-42. doi: 10.1046/j.1360-0443.2001.961217253.x. PMID 11784466
- [Background] Samet JH, Rollnick S, Barnes H. Beyond CAGE. A brief clinical approach after detection of substance abuse. Arch Intern Med. 1996 Nov 11;156(20):2287-93. doi: 10.1001/archinte.156.20.2287. PMID 8911235
- [Background] Koblin B, Chesney M, Coates T; EXPLORE Study Team. Effects of a behavioural intervention to reduce acquisition of HIV infection among men who have sex with men: the EXPLORE randomised controlled study. Lancet. 2004 Jul 3-9;364(9428):41-50. doi: 10.1016/S0140-6736(04)16588-4. PMID 15234855
- [Background] Macalino GE, Celentano DD, Latkin C, Strathdee SA, Vlahov D. Risk behaviors by audio computer-assisted self-interviews among HIV-seropositive and HIV-seronegative injection drug users. AIDS Educ Prev. 2002 Oct;14(5):367-78. doi: 10.1521/aeap.14.6.367.24075. PMID 12413183
- [Background] Delucchi KL, Jones RT, Batki SL. Measurement properties of quantitative urine benzoylecgonine in clinical trials research. Addiction. 1997 Mar;92(3):297-302. PMID 9219391
- [Background] Batki SL, Washburn AM, Delucchi K, Jones RT. A controlled trial of fluoxetine in crack cocaine dependence. Drug Alcohol Depend. 1996 Jun;41(2):137-42. doi: 10.1016/0376-8716(96)01233-1. PMID 8809502
- [Background] Preston KL, Epstein DH, Cone EJ, Wtsadik AT, Huestis MA, Moolchan ET. Urinary elimination of cocaine metabolites in chronic cocaine users during cessation. J Anal Toxicol. 2002 Oct;26(7):393-400. doi: 10.1093/jat/26.7.393. PMID 12422991
- [Background] Sobell LC, Brown J, Leo GI, Sobell MB. The reliability of the Alcohol Timeline Followback when administered by telephone and by computer. Drug Alcohol Depend. 1996 Sep;42(1):49-54. doi: 10.1016/0376-8716(96)01263-x. PMID 8889403
- [Background] Tziortzis D, Mahoney JJ 3rd, Kalechstein AD, Newton TF, De La Garza R 2nd. The relationship between impulsivity and craving in cocaine- and methamphetamine-dependent volunteers. Pharmacol Biochem Behav. 2011 Apr;98(2):196-202. doi: 10.1016/j.pbb.2010.12.022. Epub 2011 Jan 6. PMID 21215769
- [Background] Gonzalez-Saiz F, Domingo-Salvany A, Barrio G, Sanchez-Niubo A, Brugal MT, de la Fuente L, Alonso J. Severity of dependence scale as a diagnostic tool for heroin and cocaine dependence. Eur Addict Res. 2009;15(2):87-93. doi: 10.1159/000189787. Epub 2009 Jan 10. PMID 19142008
- [Background] Hunt MK, Hopko DR, Bare R, Lejuez CW, Robinson EV. Construct validity of the Balloon Analog Risk Task (BART): associations with psychopathy and impulsivity. Assessment. 2005 Dec;12(4):416-28. doi: 10.1177/1073191105278740. PMID 16244122
- [Background] Reise SP, Moore TM, Sabb FW, Brown AK, London ED. The Barratt Impulsiveness Scale-11: reassessment of its structure in a community sample. Psychol Assess. 2013 Jun;25(2):631-42. doi: 10.1037/a0032161. Epub 2013 Apr 1. PMID 23544402
- [Background] McCann DJ, Li SH. A novel, nonbinary evaluation of success and failure reveals bupropion efficacy versus methamphetamine dependence: reanalysis of a multisite trial. CNS Neurosci Ther. 2012 May;18(5):414-8. doi: 10.1111/j.1755-5949.2011.00263.x. Epub 2011 Oct 18. PMID 22070720
- [Background] Day SJ, Altman DG. Statistics notes: blinding in clinical trials and other studies. BMJ. 2000 Aug 19-26;321(7259):504. doi: 10.1136/bmj.321.7259.504. No abstract available. PMID 10948038
- [Background] Lash TL, Ahern TP. Bias analysis to guide new data collection. Int J Biostat. 2012 Jan 6;8(2):/j/ijb.2012.8.issue-2/1557-4679.1345/1557-4679.1345.xml. doi: 10.2202/1557-4679.1345. PMID 22499734
- [Background] Negus SS, Banks ML. Learning from lorcaserin: lessons from the negative clinical trial of lorcaserin to treat cocaine use disorder. Neuropsychopharmacology. 2020 Nov;45(12):1967-1973. doi: 10.1038/s41386-020-00815-4. Epub 2020 Aug 24. No abstract available. PMID 32839526
- [Background] Palacios JM, Pazos A, Hoyer D. A short history of the 5-HT2C receptor: from the choroid plexus to depression, obesity and addiction treatment. Psychopharmacology (Berl). 2017 May;234(9-10):1395-1418. doi: 10.1007/s00213-017-4545-5. Epub 2017 Mar 7. PMID 28265714
- [Background] Li SH, Chiang CN, Tai BC, Marschke CK, Hawks RL. Quantitative versus qualitative urinalysis for benzoylecgonine in clinical trials for the assessment of cocaine use. Psychopharmacol Bull. 1995;31(4):671-9. PMID 8851639
- [Result] Santos GM, Ikeda J, Coffin P, Walker JE, Matheson T, McLaughlin M, Jain J, Vittinghoff E, Batki SL. Pilot study of extended-release lorcaserin for cocaine use disorder among men who have sex with men: A double-blind, placebo-controlled randomized trial. PLoS One. 2021 Jul 15;16(7):e0254724. doi: 10.1371/journal.pone.0254724. eCollection 2021. PMID 34265007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: On 2/13/2020, the Food and Drug Administration (FDA) issued a safety alert after concluding the assessment of the long-term safety of lorcaserin in CAMELLIA clinical trial among 6,000 participants who took lorcaserin for over 4.3 years and were overweight or obese, with cardiovascular disease. The analysis showed an increased risk of cancer. In response to the safety alert, active participants in our study were instructed to stop study medication use and informed of the FDA safety alert.
Groups:
- Experimental: lorcaserin, extended release
  lorcaserin: lorcaserin 20 mg tablet
- Control: Placebo
  Placebo Oral Tablet: placebo 20 mg. tablet
Period: Overall Study
Arm/Group | Experimental | Control
Started | 16 | 6
Completed | 16 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treatment and control assignments
Groups:
- Treatment: lorcaserin, extended release
  lorcaserin: lorcaserin 20 mg tablet
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 16 | 6 | 22
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [29 to 51] | 40 [39 to 62] | 39 [32 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 15 | 4 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 7 | 2 | 9
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 6 | 22
Ever Received Cocaine Treatment [Count of Participants; unit: Participants] | 6 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Weekly Follow-up Visits of Randomized Study Participants
Description: To determine the feasibility of retaining individuals on lorcaserin vs. placebo, the investigators have calculated the mean weekly percentage of follow-up visits of those randomized in the study
Time Frame: 12 weeks
Population: The Food and Drug Administration (FDA) issued an early termination of this study after concluding the assessment in the long-term safety of lorcaserin in another clinical trial among obese, cardiovascular patients who had been taking lorcaserin for an average of 4.3 years. At the time of early termination, we had enrolled a total of 22 participants and this is why the overall number varies for this analysis.
Measure: Mean (Standard Deviation); unit: mean percent of visit retention
Groups:
- Mean Percent of Weekly Follow-up Visits by Treatment and Control Arms: Weekly Retention of randomized study participants by lorcaserin and placebo arms
Arm/Group | Mean Percent of Weekly Follow-up Visits by Treatment and Control Arms
Number analyzed (Participants) | 22
mean percent of visit retention
  Treatment Group: number analyzed (Participants) | 16
  Treatment Group | 83 (22)
  Control Group: number analyzed (Participants) | 6
  Control Group | 81 (26)
Statistical Analysis 1: Comparison: Mean Percent of Weekly Follow-up Visits by Treatment and Control Arms; Test type: Superiority; p = 0.91, Fisher Exact

2. Primary Outcome: Adverse Clinical Events in the Lorcaserin and Placebo Arms (Descriptive)
Description: To explore the tolerability of lorcaserin vs. placebo the investigators will compute the number of adverse events, both overall and by type. A participant could have more than one AE.
Time Frame: 12 weeks
Measure: Count of Units; unit: Adverse Events
Units Other Than Participants: Adverse Events
Groups:
- Treatment Group: lorcaserin, extended release
  lorcaserin: lorcaserin 20 mg tablet
- Control Group: Placebo
  Placebo Oral Tablet: placebo 20 mg. tablet
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 16 | 6
Number analyzed (Adverse Events) | 15 | 7
Adverse Events
  Hyperglycemia | 3 | 1
  Coughing | 2 | 1
  Abdominal Pain | 2 | 1
  Rash | 3 | 0
  Diarrhea | 3 | 0
  Other | 2 | 4
Statistical Analysis 1: Comparison: Treatment Group vs Control Group; Test type: Superiority; p = 0.53, Fisher Exact

3. Primary Outcome: Cumulative Percent Adherence of Medication Events Monitoring (MEMs) Cap
Description: To evaluate the adherence of lorcaserin vs. placebo, the investigators measured adherence as the frequency of taking the study drug as measured by the number of MEMS cap openings (wireless medication monitoring devices that record each opening as a real-time medication event). Cumulative percent adherence was calculated by dividing the frequency of openings at a given time point divided by the number of days since baseline.
Time Frame: 12 weeks
Population: MEMS Cap openings will track daily adherence; each dispenser opening is recorded as a medication event sent to a remote database in real time. The MEMs Cap openings will be calculated as the proportion of MEMs Cap opening over the number of days since enrollment.
Measure: Mean (Standard Deviation); unit: percent adherence
Arm/Group | Experimental | Control
Number analyzed (Participants) | 16 | 6
percent adherence | 51.6 (27.7) | 66.2 (21.7)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = .32, Fisher Exact

4. Primary Outcome: Proportion of Self-reported Past Week Cocaine Use Among Lorcaserin and Placebo Groups at Baseline and at 12 Weeks
Description: The outcome measure determines the proportion of self-reported past week cocaine use by Time-Line-Follow-back (TLFB) among lorcaserin and placebo groups at Baseline and at 12 weeks.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 16 | 6
Participants
  Proportion of self-reported weekly cocaine use by Time-Line-Follow-Up (TLFU) at baseline | 12 | 6
  Proportion of self-reported weekly cocaine use by TLFU at Week 12: number analyzed (Participants) | 13 | 6
  Proportion of self-reported weekly cocaine use by TLFU at Week 12 | 7 | 6
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = .541, Fisher Exact

5. Primary Outcome: Proportion of Urine-positive Samples With Cocaine Positivity Among Lorcaserin and Placebo Groups at Baseline and at Week 12
Description: The outcome measure determines the proportion of urine-positive samples with cocaine positivity among lorcaserin and placebo groups at Baseline and at Week 12
Time Frame: Week 12
Population: At baseline, we had 16 participants in the lorcaserin arm and 6 in the placebo arm. 8 participants in the lorcaserin arm and no participants in the placebo arm tested positive for cocaine use disorder cocaine use disorder (CUD). At week 12, four participants lost to follow-up (LTFU) in the lorcaserin arm and 1 LTFU in the placebo arm, thus causing a difference in the overall number analyzed at week 12.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 16 | 6
Participants
  Urine positive samples with cocaine use at baseline | 8 | 0
  Urine positive samples with cocaine use at Week 12: number analyzed (Participants) | 12 | 5
  Urine positive samples with cocaine use at Week 12 | 7 | 1
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.24 to 3.82]

ADVERSE EVENTS:
Time Frame: After baseline, Adverse event data were collected weekly over the 12 week period of the study.
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/16 | 1/6
Other Adverse Events (participants affected / at risk) | 16/16 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=16) | Control (N=6)
Plasma Alanine aminotransferase level and plasma aspartate aminotransferase levels (Hepatobiliary disorders) | 0 (0) | 1 (1) — One Severe Adverse Event (SAE) occurred with a participant from the placebo group and involved increased AST (Grade 3 AE) and increased ALT (Grade 2 AE) at month 1 of treatment (resolving to Grade 2 and Grade 1 AEs at the end of study participation).
Abscess of Hip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The other SAE was observed in a participant in the lorcaserin group who developed an abscess on his left hip that resolved after a course of antibiotics and was determined to not be related to lorcaserin.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=16) | Control (N=6)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) — Diarrhea SNOMED CT 409966000
abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) — abdominal pain in the stomach SNOMED CT 21522001
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — Hypoglycemia SNOWMED CT 302866003
Decreased appetite (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 2 (2) — Malaise and fever
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Coughing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early by the FDA due to the publication of a long-term safety study that showed an increase risk for cancer by the lorcaserin arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT03192995/Prot_SAP_002.pdf